CLINICAL TRIAL: NCT03967652
Title: Diagnosing Cancers From Healthy From Human Exhaled Breath With Na-nose
Brief Title: Cancer Diagnoses From Exhaled Breath With Na-nose
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anhui Medical University (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Hu Liu, Professor, Anhui Provincial Hospital
Other Study IDs: NanoBreathDiag
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Volatile Organic Compounds; Cancer; Diagnoses Disease
Keywords: Volatile organic chemicals; Cancer; Diagnose Disease; Na-nose; breath diagnoses
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cancer: Patients with definitively diagnosed of solid tumors
  Interventions: Diagnostic Test: Nanomaterial-based sensors
- Benign disease: Patients with definitively diagnosed of benign disease or precancerous lesion
  Interventions: Diagnostic Test: Nanomaterial-based sensors
- Normal: Healthy volunteers
  Interventions: Diagnostic Test: Nanomaterial-based sensors

INTERVENTIONS:
Diagnostic Test: Nanomaterial-based sensors — Chemical sensors based on Monolayer-Capped Metallic Nanoparticles (MCMNPs) can recognize and classify exhaled breath by special recognition algorithm, which achieves the purpose of disease diagnosis.

SUMMARY:
Early diagnoses of malignant tumors are pivotal for improving their prognoses. The Exhaled Breath is made up of oxygen, carbon dioxide, nitrogen, water, inert gases and volatile organic compounds (VOCs). Theoretically, the concentration of VOCs in exhalation produced by metabolism in human body is only about nmol/L-pmol/L, which can significantly increase under certain pathological conditions. A series of studies of VOCs diagnosing solid tumors the investigators had been conducted in the past decade. It was found that VOCs in exhaled breath can not only distinguish different types of tumors, but also can make a clear distinction between different stages. Our long-term collaborator, Professor Hossam Haick (Israel Institute of Technology) has developed a nano sensor array, so called Na-nose, which can detect VOCs of the exhaled breath by binding gases to specific chemiresistors coated with gold nanomaterials. The Na-nose has the advantages of low cost, easy to use, good reproducibility and real-time detection for large scale clinical application. This study was to use large clinical samples to validate the diagnostic efficacy of the newly developed Nano-nose( Sniffphone and Breath Screener) for malignant tumors .

DETAILED DESCRIPTION:
Israel Institute of Technology provides two type of Na-nose. One is Breath Screener used for large-scale sampling and feature VOCs extraction to establish database. The other is called Sniff Phone aim at clinical real-time VOCs detection assisted by software. About 10,000 patients will participate in the subject of Breath Screener in batches. First, 7000 patients will have a definitive diagnosis and exhaled breath collected. Feature VOCs of specific tumors will be extracted from these samples and employed to build predictive model by using discriminant factor analysis (DFA). After the predictive model had been completed, 3000 definitively diagnosed patients will participate in validating the specificity and sensitivity of the prediction model. With the assistance of Breath Screener clinical database and software services, Sniff Phone is more suitable for clinical real-time detection for its small and convenient design characteristics. At last, Breath Screener and Sniff Phone will continue enriching databases and improve diagnosis efficacy in their clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Cancer/benign disease having been diagnosed by pathology
* ECOG < 2

Exclusion Criteria:

* Concomitant malignancies other than one malignant tumor
* Diabetes, Fatty liver
* Autoimmune disease
* Ventilation and transaired function obstacle

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10,000 volunteers who had a definitively diagnosis with surgery or endoscope
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Build predictive diagnosis database | From July 01,2019 to December 31,2021
  First, feature VOCs of specific tumors will be extracted from part of collected samples and employed to build predictive model. After the predictive model had been completed, number of definitively diagnosed patients will participate in validating the specificity and sensitivity of the prediction model.

SECONDARY OUTCOMES:
Associated feature exhaled breath with differentially expressed genes | From Juan 01,2022 to December 31,2022
  Integrate the correlation and relevance between the exhaled samples and the differentially expressed genes in the cancer group and the benign / normal control group to explore the mechanism of feature VOCs' production.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Liu, MD, Principal Investigator — Anhui Provincial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakhleh MK, Amal H, Jeries R, Broza YY, Aboud M, Gharra A, Ivgi H, Khatib S, Badarneh S, Har-Shai L, Glass-Marmor L, Lejbkowicz I, Miller A, Badarny S, Winer R, Finberg J, Cohen-Kaminsky S, Perros F, Montani D, Girerd B, Garcia G, Simonneau G, Nakhoul F, Baram S, Salim R, Hakim M, Gruber M, Ronen O, Marshak T, Doweck I, Nativ O, Bahouth Z, Shi DY, Zhang W, Hua QL, Pan YY, Tao L, Liu H, Karban A, Koifman E, Rainis T, Skapars R, Sivins A, Ancans G, Liepniece-Karele I, Kikuste I, Lasina I, Tolmanis I, Johnson D, Millstone SZ, Fulton J, Wells JW, Wilf LH, Humbert M, Leja M, Peled N, Haick H. Diagnosis and Classification of 17 Diseases from 1404 Subjects via Pattern Analysis of Exhaled Molecules. ACS Nano. 2017 Jan 24;11(1):112-125. doi: 10.1021/acsnano.6b04930. Epub 2016 Dec 21. PMID 28000444
- [Background] Barash O, Zhang W, Halpern JM, Hua QL, Pan YY, Kayal H, Khoury K, Liu H, Davies MP, Haick H. Differentiation between genetic mutations of breast cancer by breath volatolomics. Oncotarget. 2015 Dec 29;6(42):44864-76. doi: 10.18632/oncotarget.6269. PMID 26540569
- [Background] Amal H, Shi DY, Ionescu R, Zhang W, Hua QL, Pan YY, Tao L, Liu H, Haick H. Assessment of ovarian cancer conditions from exhaled breath. Int J Cancer. 2015 Mar 15;136(6):E614-22. doi: 10.1002/ijc.29166. Epub 2014 Sep 5. PMID 25159530
- [Background] Amal H, Leja M, Broza YY, Tisch U, Funka K, Liepniece-Karele I, Skapars R, Xu ZQ, Liu H, Haick H. Geographical variation in the exhaled volatile organic compounds. J Breath Res. 2013 Dec;7(4):047102. doi: 10.1088/1752-7155/7/4/047102. Epub 2013 Nov 1. PMID 24184568
- [Background] Leja MA, Liu H, Haick H. Breath testing: the future for digestive cancer detection. Expert Rev Gastroenterol Hepatol. 2013 Jul;7(5):389-91. doi: 10.1586/17474124.2013.811033. No abstract available. PMID 23899275
- [Background] Amal H, Ding L, Liu BB, Tisch U, Xu ZQ, Shi DY, Zhao Y, Chen J, Sun RX, Liu H, Ye SL, Tang ZY, Haick H. The scent fingerprint of hepatocarcinoma: in-vitro metastasis prediction with volatile organic compounds (VOCs). Int J Nanomedicine. 2012;7:4135-46. doi: 10.2147/IJN.S32680. Epub 2012 Jul 30. PMID 22888249
- [Background] Xu ZQ, Broza YY, Ionsecu R, Tisch U, Ding L, Liu H, Song Q, Pan YY, Xiong FX, Gu KS, Sun GP, Chen ZD, Leja M, Haick H. A nanomaterial-based breath test for distinguishing gastric cancer from benign gastric conditions. Br J Cancer. 2013 Mar 5;108(4):941-50. doi: 10.1038/bjc.2013.44. PMID 23462808